CLINICAL TRIAL: NCT06124768
Title: Comparison Of Percutaneous Mechanical Thrombectomy With Different Access in Treatment of Acute Deep Venous Thrombosis (The CODA Study)
Brief Title: Comparison Of Percutaneous Mechanical Thrombectomy With Different Access in Treatment of Acute Deep Venous Thrombosis
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: First People's Hospital of Hangzhou (Other); Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: The CODA study
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep venous thrombosis; Percutaneous mechanical thrombectomy; Post-thrombotic syndrome
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Iliofemoral DVT with distal popliteal vein thrombosis treated by PMT through the modified access: Anterograde venography shows patients with iliofemoral DVT with distal popliteal vein thrombosis. PMT is performed via ipsilateral distal calf venous access or contralateral femoral access.
  Interventions: Procedure: Percutaneous mechanical thrombectomy (PMT) by the modified approach
- Iliofemoral DVT with distal popliteal vein thrombosis treated by PMT through the traditional access: Anterograde venography shows patients with iliofemoral DVT with distal popliteal vein thrombosis. PMT is performed via ipsilateral popliteal venous access.
  Interventions: Procedure: Percutaneous mechanical thrombectomy (PMT) by the traditional approach
- Iliofemoral DVT without distal popliteal vein thrombosis treated by PMT: Anterograde venography shows patients with iliofemoral DVT without distal popliteal vein thrombosis. PMT is performed via any access, such as ipsilateral femoral venous access or ipsilateral popliteal venous access.
  Interventions: Procedure: Traditional approach

INTERVENTIONS:
Procedure: Percutaneous mechanical thrombectomy (PMT) by the modified approach — The modified approach includes the ipsilateral calf venous access and the contralateral femoral venous access. Through contralateral femoral venous access, a hydrophilic guide wire and a catheter will be crossover through the thrombus side to the distal calf vein. The ipsilateral calf venous access will be punctured under the guidance of ascending venography. A hydrophilic guide wire and a catheter will be used to pass through the thrombus antegrade to the inferior vena cava. Percutaneous mechanical thrombectomy (PMT) catheter will be used to clear the thrombus. After PMT treatment, residual thrombus will be reevaluated by ascending venography. Catheter-directed thrombolysis (CDT) will be conducted if there is residual thrombus. Percutaneous balloon angioplasty (PTA) and stenting will be conducted if there is >50% stenosis of the diameter of the iliac vein.
  Groups: Iliofemoral DVT with distal popliteal vein thrombosis treated by PMT through the modified access
Procedure: Percutaneous mechanical thrombectomy (PMT) by the traditional approach — The traditional approach will be punctured from the ipsilateral popliteal vein under ultrasound guidance. A hydrophilic guide wire and a catheter will be used to pass through the thrombus antegrade to the inferior vena cava. Percutaneous mechanical thrombectomy (PMT) catheter will be used to clear the thrombus. After PMT treatment, residual thrombus will be reevaluated by ascending venography. Catheter-directed thrombolysis (CDT) will be conducted if there is residual thrombus. Percutaneous balloon angioplasty (PTA) and stenting will be conducted if there is >50% stenosis of the diameter of the iliac vein.
  Groups: Iliofemoral DVT with distal popliteal vein thrombosis treated by PMT through the traditional access
Procedure: Traditional approach — The approach will be punctured from either the ipsilateral femoral vein or popliteal vein. A hydrophilic guide wire and a catheter will be used to pass through the thrombus antegrade to the inferior vena cava. Percutaneous mechanical thrombectomy (PMT) catheter will be used to clear the thrombus. After PMT treatment, residual thrombus will be reevaluated by ascending venography. Catheter-directed thrombolysis (CDT) will be conducted if there is residual thrombus. Percutaneous balloon angioplasty (PTA) and stenting will be conducted if there is >50% stenosis of the diameter of the iliac vein.
  Groups: Iliofemoral DVT without distal popliteal vein thrombosis treated by PMT

SUMMARY:
The study aims to compare the modified approach through ipsilateral deep calf venous access or contralateral femoral venous access with the traditional approach through ipsilateral popliteal venous access for iliofemoral deep venous thrombosis (DVT) with distal popliteal vein thrombosis, and determine whether it can achieve similar therapeutic effects as iliofemoral DVT without distal popliteal vein thrombosis.

DETAILED DESCRIPTION:
Acute deep venous thrombosis (DVT) is associated with development of post-thrombotic syndrome (PTS). Early removal of iliofemoral thrombosis by percutaneous mechanical thrombectomy (PMT) may reduce the incidence of PTS. In general, PMT is performed through ipsilateral popliteal venous access as a traditional approach. However, the thrombosis in distal popliteal vein cannot be removed. Previous study demonstrated that the residual thrombus may decrease the efficacy of PMT. The study aims to compare the modified approach through ipsilateral deep calf venous access or contralateral femoral venous access with the traditional approach for iliofemoral DVT with distal popliteal vein thrombosis, and determine whether it can achieve similar therapeutic effects as iliofemoral DVT without distal popliteal vein thrombosis. The purpose of this study is to obtain high-level evidence for the endovascular treatment of acute DVT.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-85 years old;
2. Acute DVT occurred no more than 14 days since the onset of disease;
3. DVT treated by percutaneous mechanical thrombectomy
4. Informed consent signed by patients.

Exclusion Criteria:

1. Patients who are known to be allergic to heparin, low molecular weight heparin, or contrast agent;
2. Women during pregnancy and lactation;
3. Patients with other diseases that may cause difficulty in the study or significantly shorten the life expectancy of patients (<6 months);
4. Patients who are unable or unwilling to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute lower limb deep venous thrombosis (DVT) treated by percutaneous mechanical thrombectomy (PMT). The symptoms of DVT should no more than 14 days.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Immediate patency rate | Immediately after lonely percutaneous mechanical thrombectomy
  Percentage of patency rate immediately after lonely percutaneous mechanical thrombectomy
Incidence of post-thrombotic syndrome | 24-month
  Incidence of post-thrombotic syndrome (PTS) evaluated by Villalta score

SECONDARY OUTCOMES:
Rate of catheter-directed thrombolysis | Immediately after interventional surgery
  Percentage of catheter-directed thrombolysis after mechanical thrombectomy
Total time of interventional surgery | Immediately after interventional surgery
  Total time measured by hours of interventional surgery (Including duration of subsequent catheter directed thrombolysis)
Total dosage of urokinase | Immediately after interventional surgery
  Total dosage measured by units of urokinase used for procedure
Patency rate of lower limb vein | 24-month
  Percentage of patency rate of lower limb vein evaluated by ultrasound
Incidence of post-thrombotic syndrome | 12-month
  Incidence of post-thrombotic syndrome (PTS) evaluated by Villalta score
Re-intervention rate | 24-month
  Percentage of re-intervention rate for the same limb

CONTACTS AND LOCATIONS:
Overall Officials: Ni Qihong, M.D., Study Director — Department of Vascular Surgery, Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China